CLINICAL TRIAL: NCT04353193
Title: Hemodynamic Profile of Terlipressin and Octreotide in Patients With Cirrhosis and Portal Hypertension. A Randomised, Single Blinded Clinical Trial.
Acronym: INFUTER
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INFUTER; 2019-004328-39 (EudraCT Number)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Liver Cirrhosis Portal
MeSH Terms: interventions — Terlipressin; Octreotide

STUDY DESIGN:
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Terlipressin IV bolus (Experimental): Terlipressin 1mg IV bolus
  Interventions: Drug: Terlipressin
- Terlipressin IV continuous infusion (Experimental): Terlipressin by IV continuous infusion at a rate of 2mg/day (max 4mg/day) during 2 hours
  Interventions: Drug: Terlipressin
- Octreotide IV bolus plus continuous infusion (Experimental): Octreotide 50mcg IV bolus plus continuous infusion at a rate of 50mcg/h during 2 hours
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — Terlipressin 1mg IV bolus
  Arms: Terlipressin IV bolus
Drug: Terlipressin — Terlipressin by IV continuous infusion at a rate of 2mg/day (max 4mg/day) during 2 hours
  Arms: Terlipressin IV continuous infusion
Drug: Octreotide — Octreotide 50mcg IV bolus plus continuous infusion at a rate of 50mcg/h during 2 hours
  Arms: Octreotide IV bolus plus continuous infusion

SUMMARY:
Clinical trial to compare the effects of terlipressin and octreotide in the reduction of portal hypertension measured as hepatic venous pressure gradient (HVPG) in patients with liver cirrhosis

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old.
2. Liver Cirrhosis
3. Portal hypertension
4. Stable disease in the absence of vasoactive agents
5. Signed informed consent form

Exclusion Criteria:

* 1. Patients on medications that can prolong QT interval 2. Patients with HCC not fulfilling Milan criteria for transplant 3. Grade II-IV hepatic encephalopathy 4. GI bleeding in the last 10 days 5. Child-Pugh C above 12 points 6. Bacterial infection in the last 10 days 7. HVPG <12mmHg 8. Plasma sodium <130mmol/l 9. Serum creatinine >2mg/dl 10. Serum bilirubin >5mg/dl 11. INR>2.5 12. Uncontrolled cardiovascular disease 13. HIV infection 14. Extra hepatic malignancies 15. Heart failure NYHA Grade III/IV, COPD GOLD>2 16. Morbid obesity 17. Coronary heart disease or intestinal ischemia 18. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change in HVPG | 30 minutes, 1 hour and 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided